CLINICAL TRIAL: NCT07401849
Title: Blood Biomarkers for Early and Accurate Diagnosis of Alzheimer's Disease in Primary Care
Acronym: BEAD-PC
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 167698; 25/WS/0163 (Other: Research Ethics Committee (REC))
Record Dates: First submitted 2026-01-20; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Biomarkers / Blood; Biomarker in Early Diagnosis; Mild Cognitive Impairment (MCI)
Keywords: Alzheimer's Disease; Memory complaints; Mild Cognitive Impairment; Primary care; Blood biomarkers; Neuropsychological assessment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Cerebrospinal Fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alzheimer's disease is a degenerative condition affecting the brain and is the most common form of dementia in older adults. Dementia is currently a major healthcare issue in the UK, affecting approximately a million people. The progression of the disease varies between individuals and the early stages may be characterised by only minimal changes in memory and thinking. These changes could remain undetected as the symptoms may be mistakenly regarded as normal age-related forgetfulness. However, dementia is not part of the normal ageing process.

The underlying biological disease process of Alzheimer's is now known to start at least 20 years prior to patients showing any symptoms. A protein called amyloid starts to deposit in the brain and forms clumps referred to as 'plaques'. Another protein called tau collects inside brain cells and forms structures called 'tangles'. These biological changes can disrupt the normal functioning of brain cells and ultimately destroy them, leading to a reduction in brain volume and ability.

The aim of the BEAD-PC study is to assess whether a specific blood test in primary care can help diagnose Alzheimer's disease at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and above
* Presence of self-reported symptoms indicative of cognitive decline or concerns family members/partners indicative of cognitive decline
* Capacity to consent
* Be fluent in and able to read and write in English and have adequate hearing and visual acuity to complete the required psychometric tests.

Exclusion Criteria:

* Insufficient vision and hearing
* Prior diagnosis of ADRD. Prior diagnosis of Alzheimer's disease or related dementia (with or without evidence of pathology), through clinical diagnosis and/or as documented in their medical record
* Pre-existing diagnosis of dementia
* Incidental findings of brain pathologies on brain MRI, such as cancerous space occupying lesions and clinically significant vascular malformations and recent (within 12 months) macro-infarcts, that are, also exclusionary
* Contraindication for Lumbar Puncture
* Involvement in interventional research study within 3 months prior to screening
* For any other reason, in the opinion of the Investigator, participating in the study is not in the best interest of the patient.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients from 124 GP surgeries England.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Presence of Alzheimer-specific blood biomarkers | Day 1 (study entry)
  Amyloid and Tau protein biomarkers identified in blood sample
Presence of Alzheimer-specific Cerebrospinal Fluid (CSF) biomarkers | Follow-up visit (around 6 months after study entry)
  Amyloid and Tau protein biomarkers found in CSF

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) score | Day 1 (study entry)
  Pen-and-paper cognitive test commonly used to identify Mild Cognitive Impairment (MCI) in older adults.
CANTAB score | Day 1 (study entry)
  Online, self-completed battery of cognitive tests validated for detecting signs of AD-related cognitive decline.

CONTACTS AND LOCATIONS:
Overall Officials: Lefkos Middleton, Prof, Study Chair — Imperial College London; David Wingfield, Dr, Principal Investigator — Imperial College London